CLINICAL TRIAL: NCT04496713
Title: Pilot Study - Randomized Controlled Trial of Video and Telephone Primary Care Visits
Brief Title: Pilot Study of Video and Telephone Primary Care Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00257994
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-02

CONDITIONS: Telemedicine
Keywords: telemedicine; audio/video; telephone; primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine - Phone (No Intervention): Patients will continue with their telephone-based telemedicine visit as scheduled. There will be no change to their care. Patients will receive a survey by mail about the visit.
- Telemedicine - Audio/Video (Experimental): Patients will be given an internet-connected tablet to have their upcoming visit with their physician by audio/video. A survey can be completed on the tablet. The devices will be sent back to the research time after their single use.
  Interventions: Other: Internet-connected computer tablet

INTERVENTIONS:
Other: Internet-connected computer tablet — An internet-connected tablet provided to patient for upcoming visit with physician by audio/video which can also be used to complete a survey.
  Arms: Telemedicine - Audio/Video

SUMMARY:
The inability to access and use smartphones or camera-outfitted internet-connected devices during the COVID-19 pandemic relegates certain patients to receive audio-only telemedicine instead of audio/video-based telemedicine. The investigators are conducting a randomized controlled trial in order to characterize patient and provider attitudes towards these two modalities of care and to test the feasibility of a new model to make tablets for video-based care accessible to those who need that. The investigators hypothesize that patient and provider satisfaction will be higher with video-based telehealth when compared to phone-based telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for telephone-based visits who are doing so because of a lack of ability to conduct a video visit (i.e. no tablet/laptop; no access to internet) who live in Baltimore City

Exclusion Criteria:

* Patients with significant visual or hearing impairment
* Patients that have legal guardians or who are marked as lacking healthcare decision-making capacity
* Patients that have not selected English as their preferred language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Provider rating as assessed by the Consumer Assessment of Healthcare Providers and Systems question on provider rating | Within 2 weeks of the study visit
  Provider rating will be assessed with the Consumer Assessment of Healthcare Providers and Systems question on provider rating of 0-10; 0 being worst provider possible and 10 being best provider possible.

SECONDARY OUTCOMES:
Satisfaction with telemedicine visit for patient as assessed by a Likert scale | Within 2 weeks of the study visit
  Satisfaction with telemedicine visit for patient will be assessed with Likert-scale questions related to satisfaction.
  Satisfaction (1=strongly disagree to 5=strongly agree).
  1. In general, I was satisfied with using a video or phone call for this visit
  2. I could explain my medical problems well enough
  3. Talking to the doctor was as satisfying as talking in person
  Overall score 3 to 15 with higher scores signifying better satisfaction.
Satisfaction with telemedicine visit for provider as assessed by a Likert scale | Within 2 weeks of the study visit
  Satisfaction with telemedicine visit for provider will be assessed with Likert-scale questions related to satisfaction.
  [1=Strongly Disagree. 5=Strongly Agree].
  1. In general, I was satisfied with using telemedicine for this visit
  2. Talking to the patient was as satisfying as talking in person.
  Overall score 2 to 10 with higher scores signifying better satisfaction.
Efficacy of telemedicine visit for provider as assessed by a Likert scale | Within 2 weeks of the study visit
  Efficacy of telemedicine visit for provider will be assessed with Likert-scale questions related to efficacy.
  [1=Strongly Disagree. 5=Strongly Agree]. b. I was able to understand the patient's explanation of their medical problems well enough.
  c. In general, this telemedicine visit was effective in improving this patient's medical care d. An in-person visit would likely have provided additional clinically-relevant information e. An in-person visit would likely have led to a change in management
Provider communication as assessed by yes/no question | Within 2 weeks of the study visit
  The ability of a provider to communicate will be assessed by patients with the yes/no question of a modified version of the Consumer Assessment of Healthcare Providers and Systems questionnaire related to communication.
  Did this provider explain things in a way that was easy to understand? Yes/No
Provider listening as assessed by yes/no question | Within 2 weeks of the study visit
  Provider listening will be assessed by patients with the yes/no question of a modified version of the Consumer Assessment of Healthcare Providers and Systems questionnaire related to listening.
  Did this provider listen carefully to you? Yes/No
Provider respect as assessed by yes/no question | Within 2 weeks of the study visit
  Provider respect will be assessed by patients with the yes/no question of a modified version of the Consumer Assessment of Healthcare Providers and Systems questionnaire relating to respect.
  Did this provider show respect for what you had to say? Yes/No
Provider time spent as assessed by yes/no question | Within 2 weeks of the study visit
  Provider time spent will be assessed by patients with the yes/no question of a modified version of the Consumer Assessment of Healthcare Providers and Systems questionnaire relating to time spent during the clinical encounter.
  Did this provider spend enough time with you? Yes/No
Patient health rating as assessed by a likert scale | Within 2 weeks of the study visit
  Patient health will be assessed with Likert-scale questions related to patient health.
  In general, how would you rate your overall health?
  1. Excellent
  2. Very good
  3. Good
  4. Fair
  5. Poor
  In general, how would you rate your overall mental or emotional health?
  1. Excellent
  2. Very good
  3. Good
  4. Fair
  5. Poor
  Overall score 2 to 10 with lower scores signifying better health.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Epstein, MD, Principal Investigator — Johns Hopkins University; Casey Overby Taylor, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol and analysis plan, without any protected health information (PHI), can be shared on request via email.
Supporting Information: Study Protocol, SAP